CLINICAL TRIAL: NCT03676920
Title: Improving Treatment Cost Discussions Between Cancer Patients and Their Oncologists: Feasibility and Utilization of an Application-based Question Prompt List
Brief Title: Feasibility and Utilization of an Application-based Question Prompt List
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Lauren Hamel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-129
Record Dates: First submitted 2018-09-12; First posted 2018-09-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Financial Toxicity; Cancer; Question Prompt List
Keywords: cancer treatment cost, patient-provider communication
MeSH Terms: conditions — Financial Stress; Neoplasms

STUDY DESIGN:
Intervention Model Description: The research tests the feasibility of an application-based ("app") communication intervention designed to improve the frequency and quality of patient-oncologist treatment cost discussions during clinical interactions, and associated measures.
Masking Description: There is only one arm and patients will know they are testing the intervention. Physicians will not be told explicitly which of their patients are enrolled in the study but they may see patients with the intervention (either on an iPad or in a printed version).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): This feasibility study includes only one arm. All enrolled patients will be asked to use the intervention.
  Interventions: Behavioral: Discussions of Cost App (DISCO App)

INTERVENTIONS:
Behavioral: Discussions of Cost App (DISCO App) — The DISCO App is an app-based and patient-focused intervention designed to improve the frequency and quality of patient-oncologist treatment cost discussions. The DISCO App allows patients to provide basic demographic information (e.g., employment status, insurance status, etc), and uses that information to provide patients with an individually-tailored list of treatment cost questions they can ask their provider.
  Other Names: DISCO App

SUMMARY:
This trial studies how well an application-based question prompt list works in improving treatment cost discussion between patients with breast, prostate, lung, or colorectal cancer and their oncologists. An application-based question prompt list, called Discussion of Cost Application (DISCO App), may help to improve how patients and oncologists discuss cancer treatment costs.

DETAILED DESCRIPTION:
The overall goal of this research is to reduce financial toxicity related to the cost of cancer treatment in a diverse patient population. The research tests the feasibility of an application-based ("app") communication intervention designed to improve the frequency and quality of patient-oncologist treatment cost discussions during clinical interactions, which, in turn, should improve other short- and longer-term patient outcomes, including referrals to economic support (e.g., social work); efficacy in managing treatment cost; treatment cost distress; financial toxicity; and treatment adherence. If successful, this study will result in an evidence-based tool that can reduce financial toxicity and improve medical outcomes for a diverse patient population.

ELIGIBILITY:
Inclusion Criteria:

* Medical oncologists or radiation oncologists at KCI McLaren Detroit, McLaren Flint, McLaren Macomb and McLaren Port Huron oncology centers
* Oncologists will be eligible if they treat patients with prostate, breast, lung or colorectal cancers.
* Oncologists will be consented
* Patients must be 18 yrs. old or older
* Patients will be consented
* Patients must be able to read and write in English
* Patients must have a confirmed diagnosis of breast, prostate, lung or colorectal cancer and are scheduled to see an oncologist for an initial treatment discussion.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Patient-oncologist treatment cost discussions | During the treatment discussions and observed via video recordings of those discussions.
  Observational measures using video-recorded patient-oncologist treatment discussions
Patient-oncologist treatment cost discussions | Collected immediately after the interaction with the oncologist
  Self-report measures of if and how patients and oncologists discuss treatment cost.

SECONDARY OUTCOMES:
Patient financial demographics | Collected immediately prior to the interaction with the oncologist
  Patient financial situation (e.g., income, perceived economic burden, etc.)
Change in patient treatment cost information desired and gained | Collected immediately prior to and immediately after the interaction with the oncologist
  What cost treatment information patients want before the interaction and if they gained it during the interaction with their oncologist.
Change in patient efficacy in managing treatment cost (10-item scale). This measure will assess any change in the patients' efficacy in paying for the cost of their cancer treatment before and after the intervention. | Collected immediately prior to and immediately after the interaction with the oncologist
  If patients think they will be able to pay for the cost of their cancer treatment. This is adapted from a validated 10-item scale (Peterson AM, Harper FW, Albrecht TL, et al. Parent caregiver self-efficacy and child reactions to pediatric cancer treatment procedures. J Pediatr Oncol Nurs. 2014;31(1):18-27.) An example item is: "I am confident I can pay for the costs of my treatment." Patients will respond to a scale from Strongly Disagree (1) to Strongly Agree (5) with higher values representing a better outcome.
Satisfaction with treatment cost discussions (3-item scale). This will assess the extent to which patients are satisfied with any discussions of treatment cost they had with their oncologist. | Collected immediately after the interaction with the oncologist
  The extent to which patients are satisfied with any treatment cost discussion they had with their oncologist. This is an investigator-developed 3-item scale. An example item is: "I am satisfied with how my oncologist and I discussed treatment cost today." Patients will respond to a scale from Strongly Disagree (1) to Strongly Agree (5) with higher values representing a better outcome.
Length of the interaction | During the patient-oncologist interaction and observed via video recordings of the treatment discussions
  Observer measure of the length of the patient-oncologist collected using video recordings.
DISCO App use (observer measure) | Prior to and during the patient-oncologist interaction
  Observer measure of how patients use the DISCO App collected using video recordings

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Hamel, Ph.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Derived] Hamel LM, Dougherty DW, Hastert TA, Seymour EK, Kim S, Assad H, Phalore J, Soulliere R, Eggly S. The DISCO App: A pilot test of a multi-level intervention to reduce the financial burden of cancer through improved cost communication. PEC Innov. 2021 Oct 30;1:100002. doi: 10.1016/j.pecinn.2021.100002. eCollection 2022 Dec. PMID 37364004